CLINICAL TRIAL: NCT03154034
Title: Cardiopulmonary Exercise Testing in Severe Mitral Regurgitation - a Single Center, Observational Echocardiographic Study
Brief Title: Cardiopulmonary Exercise Testing in Severe Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Dr. Alexander Dietl, Resident, University Hospital Regensburg
Other Study IDs: UHRegensburg1
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Mitral Valve Regurgitation; Pulmonary Hypertension
Keywords: Stress echocardiography; Cardiopulmonary exercise testing; ergospirometry
MeSH Terms: conditions — Mitral Valve Insufficiency; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood (serum and plasma samples)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe mitral regurgitation

SUMMARY:
The purpose of this study is the evaluation of cardiac and pulmonary response to cardiopulmonary exercise in severe mitral regurgitation and its variation under treatment (surgical mitral valve repair, percutaneous mitral valve repair, optimal medical treatment). The study is conducted as a prospective, observational, single-center study. Patients suffering from symptomatic severe mitral regurgitation will be eligible, if they are referred to the University Hospital of Regensburg, Germany, for further diagnostic procedures and heart team discussion. Cardiopulmonary exercise testing is performed comprising standardized stress echocardiography as well as ergospirometry. Additional detailed assessment will be conducted including standardized questionary, clinical examination, transesophageal echocardiography and measurement of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic, severe mitral regurgitation
* referral for diagnostic work-up and heart team discussion
* declaration of informed consent

Exclusion Criteria:

* contra-indication for cardiopulmonary stress examination (unstable angina pectoris, left main disease, abnormal electrolyte concentrations, acute decompensation)
* pregnancy
* exercise test on treadmill not possible (amputation of lower extremity, severe arthritis of lower extremities)
* no acceptable acoustic window at rest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic, severe mitral regurgitation. Aetiology and treatment of mitral regurgitation do not affect enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
exercise-induced systolic pulmonary arterial pressure | Change from Baseline Exercise-Induced Systolic Pulmonary Arterial Pressure at 1 year
  exercise-induced systolic pulmonary arterial pressure measured by stress- echocardiography

SECONDARY OUTCOMES:
peak oxygen uptake (peakVO2) | Change from Baseline peakVO2 at 1 year
  peak oxygen uptake measured by ergospirometry

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dietl, MD, Principal Investigator — University Hospital Regensburg
Locations (1):
- University Hospital Regensburg - Department of Internal Medicine II, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No